CLINICAL TRIAL: NCT04482517
Title: Reproductive Outcomes of Different Sperm Selection Techniques; Density Gradient Centrifugation, Testicular Sperm, PICSI, and MACS for ICSI Patients With Abnormal Sperm DNA Fragmentation
Brief Title: Reproductive Outcomes of Different Sperm Selection Techniques for ICSI Patients With Abnormal Sperm DNA Fragmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH-005
Record Dates: First submitted 2020-07-18; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Infertility, Male
Keywords: Sperm DNA fragmentation; PICSI; MACS; Sperm Selection; DGC
MeSH Terms: conditions — Infertility, Male | interventions — Centrifugation, Density Gradient; Sperm Retrieval

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Density Gradient Centrifugation (DGC) (Other): Using the routine DGC sperm processing only
  Interventions: Other: Density Gradient Centrifugation
- Physiological ICSI (PICSI) (Active Comparator): Using PICSI dish for selecting sperm with lower sperm DNA fragmentation
  Interventions: Other: Physiological ICSI
- Magnetic Activated Cell Sorting (MACS) (Active Comparator): Using MACS for selecting sperm with lower sperm DNA fragmentation
  Interventions: Other: Magnetic activated cell sorting
- Testicular sperm (Testi) (Active Comparator): Using testicular sperm not ejaculated sperm
  Interventions: Other: Testicular sperm

INTERVENTIONS:
Other: Density Gradient Centrifugation — Semen processing is done by double layer density gradient method.
  Other Names: DGC
  Arms: Density Gradient Centrifugation (DGC)
Other: Physiological ICSI — Sperm selection by PICSI dishes depending on hyaluronan binding of sperm head
  Other Names: PICSI
  Arms: Physiological ICSI (PICSI)
Other: Magnetic activated cell sorting — Sperm selection by using Annexin V micro-beads and separation columns
  Other Names: MACS
  Arms: Magnetic Activated Cell Sorting (MACS)
Other: Testicular sperm — Using testicular sperm retrieved by TESA or TESE
  Other Names: Testi
  Arms: Testicular sperm (Testi)

SUMMARY:
Comparing the reproductive outcomes of different sperm selection techniques; Density gradient centrifugation (DGC), Testicular sperm (Testi), Physiological ICSI (PICSI), and Magnetic activated cell sorting (MACS) in abnormal sperm DNA fragmentation (SDF) ICSI patients.

ELIGIBILITY:
Inclusion Criteria:

* Female age was ≤37 years
* Female should has 5≥ metaphase II oocytes
* Males having abnormal SDF levels ≥ 20.3% by TUNEL assay
* Abstinence from 1 to 2 days
* Males having at least 1 million total motile progressive count

Exclusion Criteria:

* Leukocytospermia
* Presence of varicocele.
* Known genetic abnormality
* Use of sperm donation or cryopreserved sperm
* Use of Oocyte donation
* Use of gestational carrier
* Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previous uterine infection
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 320 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 14 days following embryo transfer
  Defined as clinical pregnancy per transfer
Implantation rate | 6- 8 weeks following embryo transfer
  Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 6 over number of embryo transferred.
Ongoing pregnancy rate | 20 weeks of gestation
  Defined as the proportion of pregnancies that completed more than 20 weeks of gestation

SECONDARY OUTCOMES:
Cleavage rate | 3 days
  Defined as the proportion of cleaved embryos on day 3 over the injected oocytes
Blastulation rate | 5-6 days
  Defined as the proportion of blastocysts formed on day 5 or 6 over the cleaved embryos on day 3
High quality blastocyst rate | 5-6 days
  Defined as the assessment of blastocyst quality according to Gardner's criteria into: good, fair or bad in terms of percentage of the total formed blastocysts
Miscarriage rate | 20 weeks of gestation
  Defined as the proportion of miscarried cases

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hasanen, Principal Investigator — Ganin Fertility Center; khaled Elqusi, Principal Investigator — Ganin Fertility Center; Salma Eltanbouly, Principal Investigator — Ganin Fertility Center; Samar Gamal, Principal Investigator — Ganin Fertility Center; Abd ElGhafar Hussin, Principal Investigator — Ganin Fertility Center; Hanaa Elkhadr, Principal Investigator — Ganin Fertility Center; Hosam Zaki, Study Chair — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Maadi, Egypt

REFERENCES:
- [Derived] Hozyen M, Hasanen E, Elqusi K, ElTanbouly S, Gamal S, Hussin AG, AlKhader H, Zaki H. Reproductive Outcomes of Different Sperm Selection Techniques for ICSI Patients with Abnormal Sperm DNA Fragmentation: a Randomized Controlled Trial. Reprod Sci. 2022 Jan;29(1):220-228. doi: 10.1007/s43032-021-00642-y. Epub 2021 Jun 2. PMID 34076869